CLINICAL TRIAL: NCT04246125
Title: Evaluation of the Patient Skin Dose in Interventional Radiology
Brief Title: Patient Skin Dose in Interventional Radiology
Acronym: DPPRI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191082; 2019-A02411-56 (Other: IDRCB)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Aneurysm; Arteriovenous Malformations; Coronary Occlusion; Lung Neoplasms; Liver Neoplasms
Keywords: Dose archiving and communication systems; Dosimetry; Gafchromic film; Interventional radiology; Peak skin dose
MeSH Terms: conditions — Aneurysm; Arteriovenous Malformations; Coronary Occlusion; Lung Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Therapeutic interventional radiology: Patients undergoing an interventional radiology procedure, at risk for developing radiation-induced skin lesions, including acts of therapeutic interventional neuroradiology (angioplasties, embolization of aneurysms, embolization of arteriovenous malformations , etc…), embolizations and ablations of thoracic tumors, therapeutic cardiac acts (transluminal angioplasties and chronic coronary occlusions) and abdominal embolizations.
  Interventions: Procedure: Interventional radiology : skin dose measurements

INTERVENTIONS:
Procedure: Interventional radiology : skin dose measurements — Therapeutic interventional radiology procedure for the following anatomical regions:
  * cerebral (neuroradiology)
  * thoracic (cardiology, lungs)
  * abdominal
  Assessment of peak skin dose and dose mapping with use of Gafchromic film dosimeter and the estimation of the absorbed dose to the skin with use of RDM software program.

SUMMARY:
Studies on radiation induced patients' skin lesions in interventional radiology highlighted the need for optimized and personalized patient dosimetry and adapted patient follow-up. Measurements using Gafchromic® films or thermoluminescent dosimeters have long been the only way to accurately evaluate the maximum absorbed dose to the patient skin. However as these dose measurements are tedious and expensive, they could not be systematically applicable in clinical practice. Therefore, more practical calculation methods have been developed. These software programs calculate the skin dose using dosimetric information from images DICOM header or radiation dose structured reports (RDSRs). Validation studies of these software programs are rare and when existent have many limitations.

Radiation Dose Monitor (RDM from Medsquare) is a software program for archiving and monitoring of radiation dose (DACS, Dosimetry Archiving Communication System) used in routine in the investigator's hospitals. A new functionality developed in RDM allows quick estimation without in-vivo measurements of the absorbed dose to the skin of the patient. Comparing RDM calculations with in-vivo measurements will enable this software validation so that it can be used in clinical routine.

Main objective: to validate RDM software for calculating patient skin dose in interventional radiology.

DETAILED DESCRIPTION:
Methodology:

The study will consist of:

* Placing a rectangular dosimeter film (dimensions: 21 x 30 cm², 1mm thick) on the examination table under the sheet before installing the patient. This film is then read using a desktop scanner and specific software to determine the absorbed dose to the patient's skin. The film is not in direct contact with the patient and will not modify the standard procedure of interventional radiology.
* Collecting the weight and height of the patient
* Collecting the dosimetric information indicated in the dose report (RDSR) generated by the radiology equipment and automatically sent to the RDM DACS server at the end of the procedure (air kerma at the interventional reference point, dose area product, fluoroscopy time, X-ray tube, table and detector positions, field size, beam filtration, high voltage kV and mA current). This data is currently archived in a regulatory way, without modifying the usual patients' care pathway. This dosimetric information in addition to the technical information related to the equipment (radiology equipment brand and model, kerma calibration factor, examination table and mattress thickness) will be used as input data to the RDM software for skin dose calculations.

These last two points are realized in the classic framework of the patient care pathway and do not modify the standard procedure.

The comparison between measured and calculated absorbed dose for the validation of the calculation software will be done anonymously. The information collected does not permit the patient identification.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) who have a therapeutic interventional radiology procedure for the following anatomical regions:

  * cerebral (neuroradiology)
  * thoracic (cardiology, lungs)
  * abdominal
* Patient informed and having expressed his non-opposition to participate in the research

Exclusion Criteria:

* Patients <18 years old
* Diagnostic interventional radiology procedure
* Demented patients unable to receive information regarding their inclusion in the research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old) for whom an interventional radiology procedure is performed
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Maximum absorbed skin dose and dose distribution | Standard duration of the interventional radiology procedure carried out as part of usual care (maximum of 8 hours)
  Measurement of the maximum absorbed dose value and dose mapping by the Gafchromic® film dosimeter (in-vivo measurements within interventional radiology procedure). Comparison between measured and calculated values by the RDM software.

CONTACTS AND LOCATIONS:
Overall Officials: Lama HADID-BEURRIER, PhD, Principal Investigator — AP-HP, Lariboisière hospital; Catherine BOUCHARD, Principal Investigator — AP-HP, Cochin hospital; Bouchra HABIB GERYES, PhD, Principal Investigator — AP-HP, Necker hospital; Joëlle Ann FEGHALI, PhD, Principal Investigator — AP-HP, Bicêtre hospital
Locations (5):
- France (5):
  - AP-HP, Bicêtre Hospital, Nuclear medicine department, Le Kremlin-Bicêtre
  - AP-HP, Lariboisière Hospital, Cardiology department, Paris
  - AP-HP, Lariboisière Hospital, Neuroradiology department, Paris
  - AP-HP, Cochin Hospital, Radiology A department, Paris
  - AP-HP, Necker-Enfants Malades Hospital, Pediatric radiology department, Paris

REFERENCES:
- [Background] Food and Drug Administration (FDA). Avoidance of serious x-ray-induced skin injuries to patients during fluoroscopically-guided procedures, 1994.
- [Background] Valentin J. Avoidance of radiation injuries from medical interventional procedures. Ann ICRP. 2000;30(2):7-67. doi: 10.1016/S0146-6453(01)00004-5. PMID 11459599
- [Background] Miller DL. Efforts to optimize radiation protection in interventional fluoroscopy. Health Phys. 2013 Nov;105(5):435-44. doi: 10.1097/HP.0b013e31829c355a. PMID 24077043
- [Background] Bor D, Olgar T, Toklu T, Caglan A, Onal E, Padovani R. Patient doses and dosimetric evaluations in interventional cardiology. Phys Med. 2009 Mar;25(1):31-42. doi: 10.1016/j.ejmp.2008.03.002. Epub 2008 Apr 25. PMID 18440265
- [Background] Ying CK, Kandaiya S. Patient skin dose measurements during coronary interventional procedures using Gafchromic film. J Radiol Prot. 2010 Sep;30(3):585-96. doi: 10.1088/0952-4746/30/3/012. Epub 2010 Sep 8. PMID 20826892
- [Background] Giordano C, D'Ercole L, Gobbi R, Bocchiola M, Passerini F. Coronary angiography and percutaneous transluminal coronary angioplasty procedures: Evaluation of patients' maximum skin dose using Gafchromic films and a comparison of local levels with reference levels proposed in the literature. Phys Med. 2010 Oct;26(4):224-32. doi: 10.1016/j.ejmp.2010.01.001. Epub 2010 Feb 8. PMID 20117030
- [Background] den Boer A, de Feijter PJ, Serruys PW, Roelandt JR. Real-time quantification and display of skin radiation during coronary angiography and intervention. Circulation. 2001 Oct 9;104(15):1779-84. doi: 10.1161/hc4001.097057. PMID 11591614
- [Background] Balter S. Methods for measuring fluoroscopic skin dose. Pediatr Radiol. 2006 Sep;36 Suppl 2(Suppl 2):136-40. doi: 10.1007/s00247-006-0193-3. PMID 16862416
- [Background] Chida K, Kagaya Y, Saito H, Takai Y, Takahashi S, Yamada S, Kohzuki M, Zuguchi M. Total entrance skin dose: an effective indicator of maximum radiation dose to the skin during percutaneous coronary intervention. AJR Am J Roentgenol. 2007 Oct;189(4):W224-7. doi: 10.2214/AJR.07.2422. PMID 17885036
- [Background] Khodadadegan Y, Zhang M, Pavlicek W, Paden RG, Chong B, Schueler BA, Fetterly KA, Langer SG, Wu T. Automatic monitoring of localized skin dose with fluoroscopic and interventional procedures. J Digit Imaging. 2011 Aug;24(4):626-39. doi: 10.1007/s10278-010-9320-7. PMID 20706859
- [Background] Sanchez RM, Vano E, Fernandez JM, Escaned J. Evaluation of a real-time display for skin dose map in cardiac catheterisation procedures. Radiat Prot Dosimetry. 2015 Jul;165(1-4):240-3. doi: 10.1093/rpd/ncv033. Epub 2015 Mar 18. PMID 25788618
- [Background] Digital Imaging and Communications in Medicine (DICOM). Supplement 94: Diagnostic X-Ray radiation Dose Reporting (Dose SR), 2005.
- [Background] 1IEC/PAS 61910-1. Medical electrical equipment - Radiation dose documentation - Part 1: Radiation dose structured report for radiography and radioscopy, 2007.
- [Background] IEC/PAS 61910-1. Medical electrical equipment - Radiation dose documentation - Part 1: Radiation dose structured report for radiography and radioscopy, 2014.
- [Background] Johnson PB, Borrego D, Balter S, Johnson K, Siragusa D, Bolch WE. Skin dose mapping for fluoroscopically guided interventions. Med Phys. 2011 Oct;38(10):5490-9. doi: 10.1118/1.3633935. PMID 21992367
- [Background] Khodadadegan Y, Zhang M, Pavlicek W, Paden RG, Chong B, Huettl EA, Schueler BA, Fetterly KA, Langer SG, Wu T. Validation and initial clinical use of automatic peak skin dose localization with fluoroscopic and interventional procedures. Radiology. 2013 Jan;266(1):246-55. doi: 10.1148/radiol.12112295. Epub 2012 Nov 9. PMID 23143024
- [Background] Bordier C, Klausz R, Desponds L. Patient dose map indications on interventional X-ray systems and validation with Gafchromic XR-RV3 film. Radiat Prot Dosimetry. 2015 Feb;163(3):306-18. doi: 10.1093/rpd/ncu181. Epub 2014 Jun 17. PMID 24939865
- [Background] Bednarek DR, Barbarits J, Rana VK, Nagaraja SP, Josan MS, Rudin S. Verification of the performance accuracy of a real-time skin-dose tracking system for interventional fluoroscopic procedures. Proc SPIE Int Soc Opt Eng. 2011 Feb 13;7961(796127):796127_1. doi: 10.1117/12.877677. PMID 21731400
- [Background] Rana VK, Rudin S, Bednarek DR. A tracking system to calculate patient skin dose in real-time during neurointerventional procedures using a biplane x-ray imaging system. Med Phys. 2016 Sep;43(9):5131. doi: 10.1118/1.4960368. PMID 27587043
- [Background] Greffier J, Van Ngoc Ty C, Bonniaud G, Moliner G, Ledermann B, Schmutz L, Cornillet L, Cayla G, Beregi JP, Pereira F. Assessment of peak skin dose in interventional cardiology: A comparison between Gafchromic film and dosimetric software em.dose. Phys Med. 2017 Jun;38:16-22. doi: 10.1016/j.ejmp.2017.05.044. Epub 2017 May 8. PMID 28610693
- [Background] Magnier F, Poulin M, Van Ngoc Ty C, Osmond E, Bonniaud G, Coulot J, Pereira B, Boyer L, Guersen J, Cassagnes L. Comparison of Patient Skin Dose Evaluated Using Radiochromic Film and Dose Calculation Software. Cardiovasc Intervent Radiol. 2018 May;41(5):762-771. doi: 10.1007/s00270-018-1888-1. Epub 2018 Feb 7. PMID 29417266
- [Background] Jones AK, Pasciak AS. Calculating the peak skin dose resulting from fluoroscopically guided interventions. Part I: Methods. J Appl Clin Med Phys. 2011 Nov 15;12(4):3670. doi: 10.1120/jacmp.v12i4.3670. PMID 22089023
- [Background] Benmakhlouf H, Bouchard H, Fransson A, Andreo P. Backscatter factors and mass energy-absorption coefficient ratios for diagnostic radiology dosimetry. Phys Med Biol. 2011 Nov 21;56(22):7179-204. doi: 10.1088/0031-9155/56/22/012. Epub 2011 Oct 25. PMID 22024474
- [Background] Menzel HG, Clement C, DeLuca P. ICRP Publication 110. Realistic reference phantoms: an ICRP/ICRU joint effort. A report of adult reference computational phantoms. Ann ICRP. 2009;39(2):1-164. doi: 10.1016/j.icrp.2009.09.001. No abstract available. PMID 19897132
- [Background] IEC 61267. Medical Diagnostic X-ray Equipment - Radiation Conditions for Use in the Determination of Characteristics, 2005.
- [Background] Greffier J, Van Ngoc Ty C, Agelou M, Coulot J, Ledermann B, Ovtchinnikoff S, Pereira F, Beregi JP, Bonniaud G. Impact of the calibration conditions of XR-RV3 films on peak skin dose measurements in interventional radiology. Radiat Prot Dosimetry. 2017 Apr 25;174(2):207-215. doi: 10.1093/rpd/ncw116. PMID 27150522
- [Background] McCabe BP, Speidel MA, Pike TL, Van Lysel MS. Calibration of GafChromic XR-RV3 radiochromic film for skin dose measurement using standardized x-ray spectra and a commercial flatbed scanner. Med Phys. 2011 Apr;38(4):1919-30. doi: 10.1118/1.3560422. PMID 21626925
- [Background] Farah J, Trianni A, Ciraj-Bjelac O, Clairand I, De Angelis C, Delle Canne S, Hadid L, Huet C, Jarvinen H, Negri A, Novak L, Pinto M, Siiskonen T, Waryn MJ, Knezevic Z. Characterization of XR-RV3 GafChromic((R)) films in standard laboratory and in clinical conditions and means to evaluate uncertainties and reduce errors. Med Phys. 2015 Jul;42(7):4211-26. doi: 10.1118/1.4922132. PMID 26133620
- [Background] Miyake Et Al H. [Medical electrical equipment - part 2-43: particular requirements for the basic safety and essential performance of X-ray equipment for interventional procedures]. Nihon Hoshasen Gijutsu Gakkai Zasshi. 2011;67(3):298-301. doi: 10.6009/jjrt.67.298. No abstract available. Japanese. PMID 21471688